CLINICAL TRIAL: NCT06214832
Title: An Observation Study on the Identification of Prescription Patterns of Lodient Tab(Telmisartan/S-amlodipine) and the Changes of Symptoms According to the Treatment Effect of Hypertension for Korean Hypertensive Patients
Brief Title: An Observation Study on the Identification of Prescription Patterns of Lodient Tab(Telmisartan/S-amlodipine)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HL-LDNT-401
Record Dates: First submitted 2024-01-03; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study identify prescription patterns of Lodient Tab and evaluate the changes of the hypertension symptoms (BP pressure) who are first prescribed and taking Lodient Tab.

DETAILED DESCRIPTION:
This study aims to observe changes in symptoms according to the treatment effect of hypertension for 6 months after Lodient Tab prescription.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 years of age
2. A person diagnosed with hypertension
3. A person who has been first prescribed Lodient Tab within the past 4 months as of the IRB approval date or is scheduled to be prescribed Lodient Tab
4. A person who voluntarily agreed in writing to this study

Exclusion Criteria:

1. Pregnant women or nursing mothers
2. Persons subject to prohibition according to the permission of the Lodient Tab
3. Patients who in the judgement of the investigator, were inappropriate to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Prescribed Lodient Tab for Hypertension Treatment
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who met target systolic blood pressure (less than 140mmHg) at 6 months of prescription for Lodient Tab compared to baseline | at 6 months of prescription for Lodient Tab compared to baseline
  The percentage of patients who met target systolic blood pressure (less than 140mmHg) at 6 months of prescription for Lodient Tab compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Minseob Song, Study Chair — Seoul song clinic
Locations (1):
- Seoul song clinic, Seoul, South Korea